CLINICAL TRIAL: NCT00679133
Title: Open-Label Dose-Escalation Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Oral MGCD265 Administered With Interruption to Subjects With Advanced Malignancies
Brief Title: Safety Study of Oral MGCD265 Administered With Interruption to Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 265-102
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Malignancies
Keywords: c-Met; VEGFR; Ron; Cancer; Tumor; Safety; Phase 1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MGCD265

INTERVENTIONS:
Drug: MGCD265 — Oral daily administration; 7 days on / 7 days off

SUMMARY:
In this study, MGCD265, a new anticancer drug under investigation, is given daily on a 7 days on / 7 days off schedule to patients with advanced malignancies to study its safety profile.

DETAILED DESCRIPTION:
MGCD265 belongs to a new class of drugs with anticancer potential, known as tyrosine kinase inhibitors. MGCD265 was shown to slow down the growth of human cancer cells in mice. Clinical studies are being pursued to evaluate the safety of MGCD265 in cancer patients.

In this study, oral MGCD265 is administered daily on a 7 days on / 7 days off schedule to patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced metastatic or unresectable malignancy that is refractory to standard therapy and/or existing therapies are not likely to achieve clinical benefit. The patient's disease must be histologically confirmed;
* Evaluable disease;
* Last dose of prior chemotherapy, radiation therapy, or investigational agents occurred at least 4 weeks before the start of therapy on Cycle 1 Day 1;
* Recovery from the adverse effects of prior therapy at the time of enrollment to ≤ grade 1 (excluding alopecia);
* Age ≥ 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2;
* Life expectancy greater than 3 months following study entry;
* Adequate renal function;
* Adequate hepatic parameters;
* Adequate bone marrow function;
* A negative serum pregnancy test at screening for women of childbearing potential (WOCBP);
* Agreement by WOCBP or men whose sexual partners are WOCBP to use two methods of adequate contraception hormonal and barrier method) prior to study entry and for the duration of the study. WOCBP and men whose sexual partners are WOCBP must continue to use two methods of contraception for 28 days and 90 days, respectively, after the last dose of study medication;
* Ability to understand and willingness to sign a written informed consent document;
* Willingness and ability to comply with study visits and activities to be performed only at the study center; and
* For the Expanded MTD Cohort, the subject must have tumors that are accessible to biopsy.

Exclusion Criteria:

* Subjects with uncontrolled concurrent illness;
* Subjects with a history of a cardiovascular illness;
* Subjects with QTc > 470 msec (including subjects on medication);
* Subjects with left ventricular ejection fraction (LVEF) < 50%;
* Subjects with leukemias or myelodysplastic syndrome;
* Immunocompromised subjects;
* Subjects with a history of autologous bone marrow transplant (BMT) within the previous five years, or subjects with organ transplants or allogeneic BMT;
* Subjects with lung tumor lesions with increased likelihood of bleeding, including: history of hemoptysis; evidence of cavitation; and invasion of aorta or pulmonary arteries by the tumor;
* Subjects with a history of brain metastasis or leptomeningeal disease; subjects with tumors likely to metastasize to the brain should have a scan performed within 2 months of start of study to rule out brain metastasis (for example breast, lung, melanoma, sarcoma, etc.);
* Subjects unable to swallow oral medications or with pre-existing gastrointestinal disorders that might interfere with proper absorption of oral drugs;
* Subjects with a history of major surgery within 28 days of first receipt of study drug;
* Nursing or pregnant women;
* Subjects with any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the opinion of the Investigator, contraindicates the use of MGCD265 Drug Product or that may render the subject at excessively high risk for treatment complications; or
* Subjects with a known hypersensitivity to any of the components of the MGCD265 Drug Product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year [Anticipated]

SECONDARY OUTCOMES:
Pharmacokinetics | 1 year [Anticipated]
Pharmacodynamics | 1 year [Anticipated]
Clinical response | 1 year [Anticipated]

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Juretic, Study Director — MethylGene Inc.
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas